CLINICAL TRIAL: NCT04669483
Title: Development, Piloting and Evaluation of an Evidence-based Informed Consent Form for Total Knee Arthroplasty
Acronym: EvAb-Pilot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other); DLR German Aerospace Center (Other)
Responsible Party: Sponsor
Other Study IDs: EvAb-P-V1
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2020-12

CONDITIONS: Consent Forms; Osteoarthritis, Knee; Arthroplasty, Replacement, Knee
Keywords: informed consent; consent form; risk communication; anxiety; nocebo effect; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group (post-interruption): Patients receive evidence-based informed consent forms for total knee arthroplasty and related anaesthesia procedures
  Interventions: Other: evidence-based informed consent form
- Control group (pre-interruption): Patients receive standard consent forms (of the study centre) for total knee arthroplasty and related anaesthesia procedures

INTERVENTIONS:
Other: evidence-based informed consent form — Evidence-based informed consent forms for total knee arthroplasty and related anesthesia procedures will be developed. The design of the evidence-based informed consent forms will be guided by an existing guideline on how to present evidence-based health information (guideline evidence-based health information) and nocebo research. The information will be presented in plain language. Benefits and harms of the procedures will be presented in absolute risk formats and in comparison with other interventions or placebo. Verbal presentations of risks lead to overestimations of risks and therefore, will not be applied exclusively. Gain and loss framing will be combined. To visualize important aspects, pictograms will be used. Information on uncertainty, missing or low quality evidence will be provided.
  Groups: Intervention group (post-interruption)

SUMMARY:
Every medical intervention requires informed consent. Informed consent may include comprehensible information about the necessity and kind of the intervention, material risks and consequences or alternative treatments. Practitioners frequently use consent forms to support the physician-patient conversation and to document informed consent. Studies show, that informed consent forms used in practice, are heterogeneous.

This study aims at investigating the effects of evidence-based informed consent forms for Total Knee Replacement and related anaesthesia procedures.

Evidence-based informed consent forms include best and latest evidence in lay language. It is hypothesized that evidence-based informed consent forms - compared to standard consent forms - improve patients' risk perception, reduce anxiety of complications and reduce the nocebo effect (unspecific negative effects caused by the way of communicating risks).

To compare evidence-based and standard informed consent forms, an Interrupted Time Series pilot study will be conducted. It is planned to include 220 patients, who are scheduled for elective total knee replacement surgery.

The accompanying qualitative analyses ensure that the (German) legal requirements for informed consent are met.

ELIGIBILITY:
Inclusion Criteria:

* Patients are scheduled for an elective total knee arthroplasty surgery
* Patients are at least 18 years old
* Patients are able to understand and speak German
* Patients are mentally competent to give consent and answer questions

Exclusion Criteria:

* Patients with revision
* Patients with posttraumatic arthrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit patients who are sheduled for an elective total knee arthroplasty surgery at the clinic for orthopedics, trauma surgery and sports traumatology of the Cologne-Merheim hospital (Germany).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Anxiety: Change from baseline anxiety after the informed consent procedure assessed by the surgical fear questionnaire and a numeric rating scale (0-10) | Anxiety will be measured at the day of consultation - approximately 4 weeks before surgery - (baseline) and one day before surgery
  The surgical fear questionnaire is a validated questionnaire for measuring patient reported fear of surgery. The questionnaire includes the following items: fear of operation, fear of anaesthesia, postoperative pain, side effects, health deterioration, failed operation, incomplete recovery, long duration of rehabilitation.
Nocebo-Effect: Proportion of patients with patient reported adverse events/complications and cummulaive number of adverse events/complications assessed by closed and open questions | approximately three days after hospital discharge
  The occurence of specific adverse events/complications (e.g. postoperative nausea and vomitting) will be queried. In addition it will be queried whether other adverse events/ complications not mentioned before have occurred.

SECONDARY OUTCOMES:
Knowledge/risk perception: Proportion of correctly answered questions assessed by knowledge questions about benefits and risks of undergoing surgery | One day before surgery
  The objective knowledge questions (e.g. correct risk assessment) will be derived when developing the evidence-based informed consent forms. The development will be based on previous experiences with the measure of informed choice.
Mean satisfaction with the physician-patient-communication and informed consent form assessed by a numeric rating scale (0-10) | One day before surgery
  Patients will be queried about their overall satisfaction with the physician-patient-communication and with the informed consent form using a numeric rating scale (0-10)
Mean Quality of life (QoL) assessed by a numeric rating scale (0-10) | approximately one month after hospital discharge
  Patients will be queried about their current overall quality of life assessed by a numeric rating scale (0-10)
Mean pain and function of the knee assessed by the Oxford Knee Score | approximately one month after hospital discharge
  The Oxford Knee Score (OKS) is a validated patient reported outcome measure for patients undergoing total knee arthroplasty, that consists of 12 questions about the individual's activities of daily live and how they have been affected by pain over the preceding four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mathes, Dr., Principal Investigator — Institute for Research in Operative Medicine (IFOM), Witten/Herdecke University
Locations (1):
- Cologne Merheim Medical Center, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Weise A, Luhnen J, Buhn S, Steffen F, Zacher S, Lauberger J, Ates DM, Bohmer A, Rosenau H, Steckelberg A, Mathes T. Development, piloting, and evaluation of an evidence-based informed consent form for total knee arthroplasty (EvAb-Pilot): a protocol for a mixed methods study. Pilot Feasibility Stud. 2021 May 13;7(1):107. doi: 10.1186/s40814-021-00843-x. PMID 33985574